CLINICAL TRIAL: NCT01184573
Title: Phase 1 Study of the Pancreatic Breath Test to Detect Early Stage Chronic Pancreatitis Utilizing the Secretin Stimulation Test
Brief Title: Novel Breath Test to Detect Early Stage Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Metabolic Solutions Inc. (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: PBT01; 1R43DK089787-01 (NIH)
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; breath test; bicarbonate
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Breath samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mild to Moderate CP: Subjects must have a history compatible with chronic pancreatitis.
- Healthy Controls: Subjects must be in good health of greater than 18 years of age.

SUMMARY:
The goal of this study is to evaluate the feasibility of using a non-invasive, non-radioactive Pancreatic Breath Test (PBT) as a diagnostic tool to detect early stages of chronic pancreatitis (CP). If successful, this method could have important advantages over existing diagnostic tests for detecting early stage CP. This diagnostic breath test may have a clinical impact if it leads to early detection of CP and intervention to mitigate disease progression.

DETAILED DESCRIPTION:
Disorders of the pancreas affect more than one million persons in this country with nearly $3 billion in health care costs. The incidence rate of chronic pancreatitis (CP) is rapidly increasing and may be related to expanded alcohol abuse. Advanced CP can be easily detected by imaging techniques. However, mild to moderate CP presents a more difficult challenge for clinicians. Imaging techniques fail to recognize less advanced CP cases about 40% of the time. The gold standard for monitoring early stage CP is the secretin stimulation test. However, the secretin stimulation test is only done in a few US centers.

The investigators have developed the Pancreatic Breath Test (PBT) as an alternative to the secretin stimulation test. The breath test uses a tracer dose of sodium 13C-bicarbonate to detect the amount of bicarbonate released after stimulation of the pancreatitis by a meal (liquid Ensure). A normal pancreas releases unlabeled bicarbonate upon stimulation, decreasing the ratio of 13C/12C of exhaled carbon dioxide. This ratio will change much less in a diseased pancreas.

A case-control study in 25 mild to moderate CP patients and 25 healthy controls will be utilized to show feasibility of the new breath test.

ELIGIBILITY:
Inclusion Criteria:

* Male of female greater than or equal to 18 years of age.
* Subjects must have the ability to give informed consent.
* Female subjects of child bearing potential must use a medically acceptable form of birth control and have a negative pregnancy test.
* For case subjects with mild to moderate chronic pancreatitis, they must have either an abnormal endoscopic ultrasound (greater than 4 abnormalities), an abnormal secretin stimulation test, an abnormal endoscopic retrograde cholangiopancreatography (ERCP), an abnormal CT scan of the pancreas (dilation of the main pancreatic duct or atrophy of the pancreas), a serum trypsin level <29 ng/ml but >20 ng/ml, or a fecal elastase of less than 200 mcg/gram stool but greater than 100 mcg/gram stool.

Exclusion Criteria:

* Females who are lactating or pregnant.
* Subjects with acute pancreatitis.
* Subjects known to have a significant medical and/or mental disease.
* Subjects receiving an investigational new drug within 30 days.
* Subjects on enzyme therapy, proton pump inhibitors, H2 receptor antagonists.
* Subjects who have had a recent febrile illness within 5 days of scheduled entry into the study. Body temperature must be normal for at least 72 hours before entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two study population groups. The case group will have evidence of mild to moderate chronic pancreatitis. The control group will be healthy without evidence of chronic disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Output of C13-CO2 | 15 minutes
  Change in C13-CO2 compared to baseline values at 5, 10, and 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Phillip P Toskes, MD, Principal Investigator — University of Florida at Gainesville; David A Wagner, PhD, Principal Investigator — Metabolic Solutions Inc.
Locations (1):
- University of Florida, Gainesville, Florida, United States